CLINICAL TRIAL: NCT06670573
Title: The Investigation of Relationship Between Allergic Rhinitis with Forward Head Posture and Anxiety in Children
Brief Title: The Relationship Between Allergic Rhinitis, Forward Head Posture, and Anxiety Levels in Iranian Children
Acronym: AR FHP Anxiety
Status: Completed | Type: Observational
Sponsor: Hormozgan University of Medical Sciences (Other)
Collaborators: Tehran University (Unknown)
Responsible Party: Principal Investigator, Mohammad Bagher Rahmati, Associate Professor, Hormozgan University of Medical Sciences
Other Study IDs: IR.UT.SPORT.REC.1403.023; Tehran University (Other: Tehran University)
Record Dates: First submitted 2024-10-29; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Forward Head Posture; Allergic Rhinitis (Disorder)
Keywords: Allergic Rhinitis; Forward Head Posture; Anxiety; Children
MeSH Terms: conditions — Rhinitis, Allergic; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 25 were healthy children: 25 were diagnosed with Allergic Rhinitis

SUMMARY:
Forward head posture is a common postural issue across all age groups, often linked to the overuse of electronic devices such as computers, smartphones, and tablets, leading to poor posture in children. Allergic rhinitis is also prevalent in children, but its effects on musculoskeletal and psychological health are not well understood.

Objective: This study aimed to explore the relationship between allergic rhinitis, forward head posture, and anxiety levels in Iranian children aged 7-12 years.

Materials and Methods: Fifty children aged 7-12 were recruited from the Allergy-Infection Clinic at Bandar Abbas Children's Hospital. The participants were divided into two groups: 25 healthy children and 25 children diagnosed with allergic rhinitis. Anxiety levels were assessed using the Spence Anxiety Scale, while forward head posture was measured by analyzing photographs of the children's body profiles using AutoCAD software.

ELIGIBILITY:
The inclusion criteria :

1. children to be between 7 to 12 years old,
2. with and without Allergic Rhinitis,
3. body mass index below 95%
4. without asthma, cardiac diseases, neuromuscular diseases, tonsillectomy, congenital anomalies,
5. using smart devices less than 3 hours.

The exclusion criteria :

1-no consent

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a randomized case- control that involved 50 children aged between 7 and 12 were enrolled in the Allergy-Infection Clinic at Bandar Abbas Children's Hospital, and the study took place between may to July 2024.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Forward Head Posture | 2 month
  Forward head posture (FHP) represents a common postural imbalance characterized by the positioning of the head in a forward orientation relative to the body's vertical axis

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Daneshmandi, Professor, Study Director — Guilan University; Mohammad Hosein Alizade, Professor, Study Director — Tehran University; Mohammad Bagher Rahmati, Associate Professor, Study Director — Hormozgan University of Medical Sciences
Locations (1):
- Tehran University, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided